CLINICAL TRIAL: NCT06240429
Title: Collagen Peptide Supplementation and Physical Exercise in Adults Over 55 Years of Age: A Randomized, Double-blind, Placebo-Controlled Clinical Trial
Brief Title: Collagen Peptide Supplementation and Physical Exercise in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CAAE 52418421.9.0000.0068
Record Dates: First submitted 2024-01-23; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Collagen Supplementation; Physical Exercise Training
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blind, placebo-controlled, 12-week clinical trial involving adults over 55 years of age. Randomization of the participants will be performed by blocks of 4 participants, which will be randomized with the help of a specific software (www.random.org/sequences/), in a ratio of 1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Supplementation (Experimental): Participants will receive a daily dose of 10 g each of collagen peptides
  Interventions: Dietary Supplement: Collagen
- Placebo (No Intervention): Participants will receive a daily dose of 10 g each of placebo

INTERVENTIONS:
Dietary Supplement: Collagen — Daily doses of 10 g collagen peptide supplementation
  Arms: Collagen Supplementation

SUMMARY:
It is known that the consumption of proteins, and their consequent hyperaminoacidemia, acts synergistically with exercise in the modulation of muscle protein synthesis. In this sense, a recent study demonstrated that supplementation of a blend of collagen and milk proteins is effective in inducing increases in muscle protein synthesis rates in combination or not with exercise. Accordingly, collagen protein supplementation has also been shown to reduce nitrogen excretion and maintain body mass in individuals undergoing caloric restriction and exercise program.

Additionally, increasing collagen peptide intake has been shown to be effective in increasing collagen synthesis and reducing musculoskeletal pain. In fact, there is evidence that collagen peptide supplementation can improve functional properties in patients with chronic ankle instability. Collagen peptides have a low molecular weight and a high proportion of proline and hydroxyproline, making them more resistant to intestinal digestion and conferring a high transport efficiency and absorption speed. Thus, collagen peptides can accumulate in connective tissue, stimulating the synthesis of extracellular matrix in chondrocytes, for example.

Taken together, the evidence suggests that collagen peptide supplementation may be potentially beneficial for improving functionality in different contexts. In this sense, global demographic projections indicate that the oldest population (>55 years old) will increase substantially in the next 50 years, surpassing 2 billion by the year 2050. Aging, which leads to loss of functionality and clinical conditions associated with muscle, bone and cartilage dysfunctions. The search for lifestyle strategies capable of ensuring quality of life and autonomy and preventing chronic diseases in older individuals is of great clinical relevance. Thus, the eventual scientific proof of the efficacy of collagen protein supplementation in this population may constitute a therapeutic alternative of broad social, marketing and clinical interest, with possible extension of benefits to other age groups and groups with other characteristics.

Thus, the present study aims to investigate whether collagen peptide supplementation combined with exercise provides gains in functionality (primary outcome), muscle mass and strength, bone remodeling markers, and quality of life in adult individuals over 55 years of age.

DETAILED DESCRIPTION:
Experimental design and ethical considerations

This is a single-center, randomized, double-blind, placebo-controlled, 12-week clinical trial involving adults over 55 years of age. All participants will be informed about the risks and benefits of participating in the study and will sign an Informed Consent Form, approved by the ethics committee.

Selected participants will be randomly allocated into two groups: collagen (COL) or placebo (PLA). Participants will receive a daily dose of 10 g each of collagen peptides or placebo. The supplements will be provided in powder form, accompanied by a standard meter, and a nutritionist who is a member of the team, blindfolded to the participant's allocation, will be responsible for the (monthly) distribution of the supplement and measurement of adherence to the protocol, through diaries containing information on the time of taking the supplement and possible complications, as well as from the receipt and weighing of the remainder in the returned jars each month.

Exercise Training Protocol

The training will be prescribed remotely, being carried out at home for the convenience of the participants. The intervention will last for 12 weeks and will include exercises to develop muscle strength, aerobic capacity, balance, and flexibility . Each session will last approximately 60 minutes. Participants should perform the exercises at home 3 times a week. The entire protocol will be individualized and always accompanied by the same coach. The control and progression of the intensity of the activity will be based on the perception of exertion reported by the participant. To this end, the Borg scale of subjective perception of exertion (RPE) will be used, segmented into: 6-8 (Very easy), 9-10 (Easy), 11-12 (Relatively easy), 13-14 (Slightly tiring), 15-16 (Tiring), 17-18 (Very tiring) and 19-20 (Exhausting).

Participants will be properly instructed about all the procedures that make up the physical training protocol beforehand when they come to the hospital complex to perform the initial evaluations. On the same day, participants will be given a diary, in which they should write down in as much detail as possible the physical activities performed in their day-to-day life, and materials containing supplementary instructions (e.g., a booklet with images and description of the exercises, and videos demonstrating their proper execution). On the days they perform the training protocol, participants should also write down additional information such as the type of exercise, intensity (degree of effort/RPE per set), number of sets completed and repetitions for each exercise performed. In the case of aerobic activities, participants must fill in the total time spent per exercise (e.g., 30 min) and the number of blocks performed (e.g., 2 blocks of 15 min).

A researcher will contact the participants weekly, on pre-scheduled days and times, to check and request information regarding the diary. At these times, the researcher will also be able to check the completed data and request additional information (e.g., adversities, challenges and barriers encountered, doubts, etc.), control the participants' adherence and establish new goals and objectives. Reported adverse events will be documented and investigated by the research team in order to monitor any risk related to the intervention.

Statistical analysis

At baseline period, the groups will be compared by independent t-test for all variables. Intra- and between-group differences for the dependent variables will be tested from mixed models for repeated measures, assuming group (placebo and collagen ) and time (before and after 12-weeks of exercise intervention) as fixed factors and subjects as random factors. In case of significant F values, analyses were performed post-hoc with Tukey adjustments. The analyses will be carried out following the principles of intention to treat. All analyses will be conducted using Statistical Analysis System software (Institute Inc., Cary, NC) and the significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* At or above 55 years of age.

Exclusion Criteria:

* use of medications that may alter muscle responses
* use of dietary supplements such as proteins, amino acids or creatine
* being on a restrictive diet
* current engagement in a strength training program
* chronic diseases such as hypertension, diabetes mellitus, heart disease, uncontrolled hypo- or hyperthyroidism
* presence of conditions that prevent participation in an exercise program.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Sit and Stand test | Before and 12-weeks of exercise training program
  sit and stand test, assessed as maximal number of stands within 30 seconds
Get up and go Test | Before and 12-weeks of exercise training program
  get up and go test, assessed as the total time to walk 20 m distance.
Maximal force production | Before and 12-weeks of exercise training program
  handgrip force, assessed as maximal kg produced.

SECONDARY OUTCOMES:
Lean body mass | Before and 12-weeks of exercise training program
  Lean body mass using dual-energy X-ray absorptiometry (lumbar spine, femur and total body) (DXA
carbox-terminal bone resorption marker telopeptide of type I collagen (CTX) | Before and 12-weeks of exercise training program
  Serum concentrations of the carbox-terminal bone resorption marker telopeptide of type I collagen (CTX) will be obtained by means of the automated electrochemiluminescence method (E411, Roche Diagnostics®, Mannheim, Germany).
N-terminal propeptide bone formation marker of type I pro-collagen (P1NP) | Before and 12-weeks of exercise training program
  Serum concentrations of N-terminal propeptide bone formation marker of type I pro-collagen (P1NP) will be obtained by means of the automated electrochemiluminescence method (E411, Roche Diagnostics®, Mannheim, Germany).
Quality of Life using the Short Form Healthy Survey | Before and 12-weeks of exercise training program
  Quality of life will be assessed using the Short Form Healthy Survey (SF-36; in portuguese version). The short-form (SF-36) yields an 8-scale profile of scores (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health). Physical component summary (primary outcome) and mental component summary were also calculated. Scores range from 0 to 100 (higher scores indicate better health quality of life).
Assessment of dietary intake - Protein | Before and 12-weeks of exercise training program
  Protein intake (total, in g; relative, in % of total energy value; relative to body weight, in g/kg/day), will be assessed before and after the intervention by means of three food diaries on non-consecutive days (including two days of the week and one day of the weekend).
Assessment of dietary intake - Carbohydrate | Before and 12-weeks of exercise training program
  Carbohydrates in the diet (total, in g; relative, in % of total energy value) will be assessed before and after the intervention by means of three food diaries on non-consecutive days (including two days of the week and one day of the weekend).
Assessment of dietary intake - Lipids | Before and 12-weeks of exercise training program
  Lipids in the diet (total, in g; relative, in % of total energy value) will be assessed before and after the intervention by means of three food diaries on non-consecutive days (including two days of the week and one day of the weekend).
Assessment of dietary intake - Total calories | Before and 12-weeks of exercise training program
  Total calories (in kcal units) will be assessed before and after the intervention by means of three food diaries on non-consecutive days (including two days of the week and one day of the weekend).
Total fat body mass | Before and 12-weeks of exercise training program
  Total fat body mass) measured using dual-energy X-ray absorptiometry (lumbar spine, femur and total body) (DXA
Areal mineral density | Before and 12-weeks of exercise training program
  Areal mineral density measured using dual-energy X-ray absorptiometry (lumbar spine, femur and total body) (DXA

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital of the School of Medicine, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No